CLINICAL TRIAL: NCT01030978
Title: Prevention of Type 2 Diabetes in Children With a Family-based Healthy Lifestyle Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0908005608; 3UL1RR024139-04S2 (NIH)
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Impaired Glucose Tolerance
Keywords: Impaired Glucose Tolerance; PreDiabetes; Diabetes Prevention
MeSH Terms: conditions — Glucose Intolerance; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family-based Healthy Lifestyle Program (Experimental): Subjects attend program with a caregiver or parent twice per week for 6 mos. Exercise is 2x/wk, behavior mod/nutrition 1 x/wk, and parent class 1 x/wk. Smart Moves curriculum is utilized for nutrition and behavior mod.
  Interventions: Behavioral: Bright Bodies Healthy Lifestyle Program
- Standard Diet & Activity Education (Control) (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Bright Bodies Healthy Lifestyle Program — Subjects attend program with a caregiver or parent twice per week for 6 mos. Exercise is 2x/wk, behavior mod/nutrition 1 x/wk, and parent class 1 x/wk. Smart Moves curriculum is utilized for nutrition and behavior mod.
  Arms: Family-based Healthy Lifestyle Program
Behavioral: Control — Subjects will be given basic instruction by clinical provider and goals will be followed up every 3 months.
  Arms: Standard Diet & Activity Education (Control)

SUMMARY:
The purpose of this study is to determine if the Bright Bodies (BB) Healthy Lifestyle Program can help reverse early abnormalities in glucose metabolism and prevent the progression to type 2 diabetes (T2DM) in high-risk, obese youth with newly-diagnosed impaired glucose tolerance (IGT).

DETAILED DESCRIPTION:
Primary Aim: (1) To determine whether youth randomized to the Bright Bodies (BB) Healthy Lifestyle Program have lower 2-hr plasma glucose levels than those randomized to standard lifestyle counseling (control) after 6 months.

Secondary Aims: (2) To determine if greater conversions from IGT to normal glucose tolerance (NGT) and less development of T2DM occurs for those in the BB vs Control Group; (3)To determine if there is improvement in anthropometric/metabolic parameters in BB vs Control Group; and (4) To determine if there is an improvement in psychosocial and family dynamic outcomes of the child in BB vs Control Group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IGT (glucose 140-199 at 2 hrs during OGTT)
* Age 11 to 16
* An interest in being enrolled in a healthy lifestyle program
* A parent/caregiver willing to participate with child in program

Exclusion Criteria:

* Psychiatric disorder or serious medical condition that would preclude participation in program
* Currently taking medication that potentially effects insulin sensitivity (eg Metformin) or causes weight gain (example: Risperidone) or weight loss (eg Xenical)
* Involvement in co-existing weight management/healthy lifestyle program
* Plans of moving out of the Greater New Haven area within six months

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
2-hour plasma glucose, category of glucose tolerance (IGT, NGT, T2DM) | 6 months

SECONDARY OUTCOMES:
Homeostasis model assessment of insulin resistance (HOMA-IR) | 6 months
Lipid profile | 6 months
Alanine aminotransferase (ALT) | 6 months
Body mass index (BMI) | 6 months
Body fat mass and % | 6 months
Blood pressure (BP) | 6 months
Piers-Harris Self-concept scale score | 6 months
Child behavior checklist score | 6 months
Family assessment device (FAD) score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Sherwin, MD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigation, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Taylor JH, Xu Y, Li F, Shaw M, Dziura J, Caprio S, Tamborlane WV, Nowicka P, Savoye M. Psychosocial predictors and moderators of weight management programme outcomes in ethnically diverse obese youth. Pediatr Obes. 2017 Dec;12(6):453-461. doi: 10.1111/ijpo.12165. Epub 2016 Jul 7. PMID 27384496